CLINICAL TRIAL: NCT07119476
Title: Does Hip Strength Impact Active Females Rate of Pelvic Floor Dysfunction?
Brief Title: Does Hip Strength Impact Active Females Rate of Pelvic Floor Dysfunction? The Primary Goal of This Research is to Collect Data on Hip Strength for Active Females and Assess if There is a Relationship Between Hip Strength and Pelvic Floor Dysfunction (PFD).
Status: Completed | Type: Observational
Sponsor: George Fox University (Other)
Responsible Party: Principal Investigator, Tess Treinen Swake, Assistant Professor of Physical Therapy, George Fox University
Other Study IDs: 2241059
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Floor Muscle Weakness; Pelvic Floor Disorder; Pelvic Pain; Hip Strength
Keywords: pelvic health; active female; pelvic floor dysfunction
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active Females: Active Females Ages 18-45

SUMMARY:
The primary goal of this research is to collect data on hip strength for active females and assess if there is a relationship between hip strength and pelvic floor dysfunction (PFD). The participants will fill out a REDCap questionnaire that includes informed consent, demographics, injury history, history of PFD and/or hip pain, characteristics of physical activity and/or sport(s), knowledge of pelvic floor musculature, and questions regarding the correlation between PFD and performance. Additionally, Patient Reported Outcomes Measurement Information System (PROMIS) surveys assessing anxiety and depression will be included. After completing the questionnaires, a one time hip strength assessment will be performed in four directions on each hip and the evaluator will be blinded to their results. Foster et al researched hip and pelvic floor strength in a different patient population (Urgency and Frequency prominent lower urinary tract symptoms) in 2021 with 18-60 year olds and did not have a classification for level of physical activity. This research group found that there was a reduction in hip external rotation and abduction strength compared to case controls. To this point, there has not been any research assessing the relationship between hip strength and relaxing versus nonrelaxing pelvic floor dysfunction and controls.

DETAILED DESCRIPTION:
Women who participate in high-level physical activity are known to have increased rates of Urinary Incontinence (UI) with prevalence rates of 28-29.6% compared to non-athletes with rates of 9.8-13.4%. The current body of research for active females in pelvic health physical therapy has focused primarily on female athletes with Urinary Incontinence (UI), which is only one symptom under the greater umbrella of Pelvic Floor Dysfunction (PFD). Likewise, systematic reviews of females with PFD have been limited to the exploration of Female UI. Pelvic Floor Dysfunction can be separated into two broad categories: relaxing and nonrelaxing. Relaxing PFD conditions are more common and include diagnoses of UI and prolapse of pelvic structures. Nonrelaxing PFD can include a broad range of non-specific symptoms. These symptoms can include voiding, anorectal, and sexual dysfunction and pain. Specifically, the pain can be insertional or deep dyspareunia, low back pain that can radiate to the thighs or groin, and pelvic pain that may be unrelated to intercourse or may occur after intercourse. Voiding issues may include a sense of incomplete emptying, bladder pain, urinary frequency, urgency or dysuria.

Research related to nonrelaxing pelvic floor dysfunction has been mostly limited to a case example, a case study related to dry needling intervention and a continuing education formatted article from Mayo Clinic. Nonrelaxing PFD has been described as a disorder where "..the muscles of the pelvic floor remain in a contracted state causing increased pressure and pain." From these articles, nonrelaxing PFD can present with a wide range of nonspecific symptoms and can negatively affect quality of life.

An additional area of interest is the impact of anxiety and depression on pelvic floor dysfunction of active females. Anxiety and depression symptoms are common in individuals with PFD (30.9% and 20.3% respectively) and athletes. High performance athletes have depression rates ranging from 6.7% to 34.0% with risk factors including female gender and playing an individual sport. In a systematic review, Beisecker et al explored depression, anxiety and stress among student athletes and found specific themes related to these symptoms, including being a female student athlete, social support, connection and interaction and health components (diet and eating patterns, sleep and alcohol use).

Foster et al researched hip and pelvic floor strength in a different patient population (Urgency and Frequency prominent lower urinary tract symptoms) in 2021 with 18-60 year olds and did not have a classification for level of physical activity. This research group found that there was a reduction in hip external rotation and abduction strength compared to case controls. To this point, there has not been any research assessing the relationship between hip strength and relaxing versus nonrelaxing pelvic floor dysfunction.

I plan to make this work public through submission to the Journal of Women's Health Physical Therapy or the Journal of Orthopaedic & Sports Physical Therapy. Additionally, I will submit my findings to the American Physical Therapy Association Combined Section Meeting for platform presentation.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-45 years
* Female gender
* Patients can either have no pelvic floor symptoms, current pelvic floor dysfunction (relaxing or nonrelaxing), or current musculoskeletal pain.
* Participants must be physically active as defined by the World Health Organization (WHO) as performing 150-300 minutes of moderate-intensity aerobic physical activity or at least 75-150 minutes of vigorous-intensity aerobic physical activity; or an equivalent combination of moderate- and vigorous-intensity activity throughout the week.

Exclusion Criteria:

* Pregnancy
* Gynecological or Obstetric Surgery within 6 months
* Active infection (including Sexually Transmitted Infection, Pelvic, Urinary Tract Infection (UTI), Yeast)
* Cancer
* Inflammatory Disease
* Connective Tissue Disease
* Or have been instructed by a Healthcare provider to not participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-45 year old females who are active as described by the WHO.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Inline Tension Dynamometer: Hip Strength Assessment | Baseline (one time assessment)
  The hip strength assessment will be performed in person and will include four strength assessments (hip abduction, hip adduction, hip external rotation and hip internal rotation) for each lower extremity.
International Consensus on Incontinence Questionnaire (ICIQ-FLUTS Long Form) | Baseline (one time assessment)
  a questionnaire that evaluates female lower urinary tract symptoms and quality of life in clinical practice and research. This questionnaire has been found to be valid, reliable, and responsive. The time required to complete this questionnaire is 4-5 minutes.
  This scale is 0-48 where all subscale scores are added and higher scores indicate greater impact of individual symptoms for the patient.
Patient Reported Outcome Measure Information System (PROMIS) | Baseline (one time assessment)
  PROMIS Anxiety- CAT that focuses on fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness).
  The scale is between 8 and 40 raw score and is converted into a t score metric and a higher score indicates greater levels of anxiety. A score of 50 represents the average and a standard deviation (SD) of 10.
  PROMIS Depression- CAT that focuses on negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose).
  The scale is between 8 and 40 raw score and is converted into a t score metric and a higher score indicates greater levels of depression. A score of 50 represents the average and a standard deviation (SD) of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- George Fox University Medical Sciences Building, Newberg, Oregon, United States

REFERENCES:
- [Background] Beisecker L, Harrison P, Josephson M, DeFreese JD. Depression, anxiety and stress among female student-athletes: a systematic review and meta-analysis. Br J Sports Med. 2024 Mar 8;58(5):278-285. doi: 10.1136/bjsports-2023-107328. PMID 38233087
- [Background] Vrijens D, Berghmans B, Nieman F, van Os J, van Koeveringe G, Leue C. Prevalence of anxiety and depressive symptoms and their association with pelvic floor dysfunctions-A cross sectional cohort study at a Pelvic Care Centre. Neurourol Urodyn. 2017 Sep;36(7):1816-1823. doi: 10.1002/nau.23186. Epub 2017 Feb 21. PMID 28220586
- [Background] Sheikhhoseini R, Arab AM. Dry Needling in myofascial tracks in Non-Relaxing Pelvic Floor Dysfunction: A case study. J Bodyw Mov Ther. 2018 Apr;22(2):337-340. doi: 10.1016/j.jbmt.2017.09.016. Epub 2017 Sep 25. PMID 29861229
- [Background] Louis-Charles K, Biggie K, Wolfinbarger A, Wilcox B, Kienstra CM. Pelvic Floor Dysfunction in the Female Athlete. Curr Sports Med Rep. 2019 Feb;18(2):49-52. doi: 10.1249/JSR.0000000000000563. PMID 30730341
- [Background] Faubion SS, Shuster LT, Bharucha AE. Recognition and management of nonrelaxing pelvic floor dysfunction. Mayo Clin Proc. 2012 Feb;87(2):187-93. doi: 10.1016/j.mayocp.2011.09.004. PMID 22305030
- [Background] Almousa S, Bandin van Loon A. The prevalence of urinary incontinence in nulliparous adolescent and middle-aged women and the associated risk factors: A systematic review. Maturitas. 2018 Jan;107:78-83. doi: 10.1016/j.maturitas.2017.10.003. Epub 2017 Oct 7. PMID 29169586
- [Background] de Mattos Lourenco TR, Matsuoka PK, Baracat EC, Haddad JM. Urinary incontinence in female athletes: a systematic review. Int Urogynecol J. 2018 Dec;29(12):1757-1763. doi: 10.1007/s00192-018-3629-z. Epub 2018 Mar 19. PMID 29552736
- [Background] Sorrigueta-Hernandez A, Padilla-Fernandez BY, Marquez-Sanchez MT, Flores-Fraile MC, Flores-Fraile J, Moreno-Pascual C, Lorenzo-Gomez A, Garcia-Cenador MB, Lorenzo-Gomez MF. Benefits of Physiotherapy on Urinary Incontinence in High-Performance Female Athletes. Meta-Analysis. J Clin Med. 2020 Oct 10;9(10):3240. doi: 10.3390/jcm9103240. PMID 33050442
- [Background] Foster SN, Spitznagle TM, Tuttle LJ, Sutcliffe S, Steger-May K, Lowder JL, Meister MR, Ghetti C, Wang J, Mueller MJ, Harris-Hayes M. Hip and Pelvic Floor Muscle Strength in Women with and without Urgency and Frequency Predominant Lower Urinary Tract Symptoms. J Womens Health Phys Therap. 2021 Jul-Sep;45(3):126-134. doi: 10.1097/jwh.0000000000000209. PMID 34366727